CLINICAL TRIAL: NCT03690804
Title: Assessment of Autonomic Co-regulation Between Newborn and Parent During Kangaroo Care Sessions in Neonatal Intensive Care Units
Acronym: Co-PAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 18CH048; 2018-A00765-50 (Other: ANSM)
Record Dates: First submitted 2018-09-24; First posted 2018-10-01 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-09

CONDITIONS: Newborn
Keywords: kangaroo care; neonatal intensive care units; autonomic co-regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- newborn is above 28 weeks of gestational age (Experimental): 40 parent-newborn duos in which the newborn is above 28 weeks of gestational age and less than 3 months of life and hospitalized in neonatal intensive care units of our university hospital (Saint-Etienne - France)
  Interventions: Device: Evaluation of Autonomic nervous system indices

INTERVENTIONS:
Device: Evaluation of Autonomic nervous system indices — The ECG signal, respiration rate, SpO2 and NIPΣ or ANI are recorded simultaneously on a computer with a capture card. The other indices of HRV will be analyzed offline: SDNN (standard deviation of all NN intervals), pNN30 (NN30 count divided by the total number of all NN intervals), pNN50 (NN50 count divided by the total number of all NN intervals), RMSSD (quadratic mean of successive R-R intervals), SD1 (standard deviation), SD2 (standard deviation), LF (low frequencies), HF (high frequencies), VLF (very low frequencies), SDANN (standard deviation of the averages of NN intervals in all 5 min segments of the entire recording), ratio LF/ HF, Ptot, Poincaré plot (plot points corresponding to each R-R space of a record).

SUMMARY:
Mother-infant separation, as a result of hospitalization, leads to stress and anxiety for both parent and infant, lowers feelings of maternal competency and corrupts bonding process.

Kangaroo Care (KC), is as a widespread procedure in which the naked newborn is placed on the parent's bare chest. KC is known to enhance neonatal outcome by improving temperature regulation, cardiorespiratory stability or psychomotor development. It also promotes mother-infant interactions and enhances parental psychological well-being.

Heart rate variability (HRV) analysis is a non-invasive tool able to consider autonomic nervous system activity. Previous studies have shown that pleasant feelings are associated with an increase of high frequencies variations index (HFnu index) reflecting a prevalence of parasympathetic activity. This one can be assess by a new monitor called NIPΣ (Neonatal index of parasympathetic activity) in newborns and ANI (Analgesic nociception index) in adults can provide a comfort index by quantifying the parasympathetic tone.

The investigators hypothesize that kangaroo care could induce an autonomic co-regulation between newborn and parent by increasing parasympathetic activity.

The study will involve 40 preterm or term newborns and their parent, performing a one hour kangaroo care session in intensive unit and neonatal intensive care unit from hospital of Saint-Etienne (France).

ELIGIBILITY:
Inclusion Criteria for the newborn :

* Neonates over 28 weeks of gestational age, under 3 months, hospitalized in neonatal intensive care units of the university hospital of Saint-Etienne (France),
* performing a one hour (or more) kangaroo care session with his parent.

Inclusion Criteria for the parent (father or mother) :

- To be a parent of a child eligible for the research protocol,

Exclusion Criteria for the newborn :

* Newborn sedated
* Newborn with a treatment known to alter the sympathetic or parasympathetic activity of the autonomic nervous system.
* Associated and severe brain pathology
* Anoxo-ischemic encephalopathy
* Unbalanced congenital heart disease,

Exclusion Criteria for the parents :

* Parent with a treatment known to alter the sympathetic or parasympathetic activity of the autonomic nervous system.
* Heart surgery or cardiac pathology
* History of psychiatric pathology

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2018-10-25 (Actual)

PRIMARY OUTCOMES:
change form baseline high frequency index (HFnu) of variability RR short-term heart rate (HRV) in the frequency domain, from the parent and the child at 1 hour | Minutes 0 (early skin to skin), 10, 20, 30, 40, 50 and 60.
  Measured during the ECG recording

SECONDARY OUTCOMES:
Evaluation of the NIPE index of comfort and discomfort (Mdoloris Medical Systems ®) for the newborn | Minutes 0 (early skin to skin), 10, 20, 30, 40, 50 and 60.
  NIPΣ (neonatal index of parasympathetic activity) : evaluate the comfort of the newborn during the skin-to-skin session.
  NIPΣ is physiologically above 60%. The threshold of discomfort in the newborn would correspond to a value <60.
Evaluation of the ANI index of comfort and discomfort (Mdoloris Medical Systems ®) for the parent. | Minutes 0 (early skin to skin), 10, 20, 30, 40, 50 and 60.
  ANI (analgesia nociception index) : evaluate an index of continuous analgesia during the skin-to-skin session.
  ANI is physiologically above 60%. The threshold of discomfort in the newborn would correspond to a value <60.
gestational age | at the inclusion
Ptot (indices of variability of heart rate) for the parent | Minutes 0 (early skin to skin), 10, 20, 30, 40, 50 and 60.
  Measured during the ECG recording
Ptot (indices of variability of heart rate) for the newborn | Minutes 0 (early skin to skin), 10, 20, 30, 40, 50 and 60.
  Measured during the ECG recording
VLF (indices of variability of heart rate) for the parent | Minutes 0 (early skin to skin), 10, 20, 30, 40, 50 and 60.
  Measured during the ECG recording
VLF (indices of variability of heart rate) for the newborn | Minutes 0 (early skin to skin), 10, 20, 30, 40, 50 and 60.
  Measured during the ECG recording
LF (indices of variability of heart rate) for the parent | Minutes 0 (early skin to skin), 10, 20, 30, 40, 50 and 60.
  Measured during the ECG recording
LF (indices of variability of heart rate) for the newborn | Minutes 0 (early skin to skin), 10, 20, 30, 40, 50 and 60.
  Measured during the ECG recording
HF (indices of variability of heart rate) for the parent | Minutes 0 (early skin to skin), 10, 20, 30, 40, 50 and 60.
  Measured during the ECG recording
HF (indices of variability of heart rate) for the newborn | Minutes 0 (early skin to skin), 10, 20, 30, 40, 50 and 60.
  Measured during the ECG recording
ratio LF/HF (indices of variability of heart rate) for the parent | Minutes 0 (early skin to skin), 10, 20, 30, 40, 50 and 60.
  Measured during the ECG recording
ratio LF/HF (indices of variability of heart rate) for the newborn | Minutes 0 (early skin to skin), 10, 20, 30, 40, 50 and 60.
  Measured during the ECG recording
SDNN (indices of variability of heart rate) for the parent | Minutes 0 (early skin to skin), 10, 20, 30, 40, 50 and 60.
  Measured during the ECG recording
SDNN (indices of variability of heart rate) for the newborn | Minutes 0 (early skin to skin), 10, 20, 30, 40, 50 and 60.
  Measured during the ECG recording
SDANN (indices of variability of heart rate) for the parent | Minutes 0 (early skin to skin), 10, 20, 30, 40, 50 and 60.
  Measured during the ECG recording
SDANN (indices of variability of heart rate) for the newborn | Minutes 0 (early skin to skin), 10, 20, 30, 40, 50 and 60.
  Measured during the ECG recording
pNN30 and pNN50 (indices of variability of heart rate) for the parent | Minutes 0 (early skin to skin), 10, 20, 30, 40, 50 and 60.
  Measured during the ECG recording
pNN30 and pNN50 (indices of variability of heart rate) for the newborn | Minutes 0 (early skin to skin), 10, 20, 30, 40, 50 and 60.
  Measured during the ECG recording
RMSSD (indices of variability of heart rate) for the parent | Minutes 0 (early skin to skin), 10, 20, 30, 40, 50 and 60.
  Measured during the ECG recording
RMSSD (indices of variability of heart rate) for the newborn | Minutes 0 (early skin to skin), 10, 20, 30, 40, 50 and 60.
  Measured during the ECG recording
SD1 and SD2 (indices of variability of heart rate) for the parent | Minutes 0 (early skin to skin), 10, 20, 30, 40, 50 and 60.
  Measured during the ECG recording
SD1 and SD2 (indices of variability of heart rate) for the newborn | Minutes 0 (early skin to skin), 10, 20, 30, 40, 50 and 60.
  Measured during the ECG recording
Poincaré-plot index (indices of variability of heart rate) for the parent | Minutes 0 (early skin to skin), 10, 20, 30, 40, 50 and 60.
  Measured during the ECG recording
Poincaré-plot index (indices of variability of heart rate) for the newborn | Minutes 0 (early skin to skin), 10, 20, 30, 40, 50 and 60.
  Measured during the ECG recording
fractal index (indices of variability of heart rate) for the parent | Minutes 0 (early skin to skin), 10, 20, 30, 40, 50 and 60.
  Measured during the ECG recording
fractal index (indices of variability of heart rate) for the newborn | Minutes 0 (early skin to skin), 10, 20, 30, 40, 50 and 60.
  Measured during the ECG recording
entropy index (indices of variability of heart rate) for the parent | Minutes 0 (early skin to skin), 10, 20, 30, 40, 50 and 60.
  Measured during the ECG recording
entropy index (indices of variability of heart rate) for the newborn | Minutes 0 (early skin to skin), 10, 20, 30, 40, 50 and 60.
  Measured during the ECG recording

CONTACTS AND LOCATIONS:
Overall Officials: Hugues PATURAL, MD PhD, Principal Investigator — CHU de Saint Etienne
Locations (1):
- CHU de Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No